CLINICAL TRIAL: NCT01568086
Title: Phase Ib Follow-up Study to Evaluate Long-term Safety and Tolerability of Immunization With AFFITOPE AD03 Applied During AFFiRiS 005A
Brief Title: Follow-up Study to Evaluate Long-term Safety and Tolerability of Immunization With AD03 Applied During AFF005A
Status: Terminated | Type: Observational
Why Stopped: The study could not be performed as planned for organizational reasons.
Sponsor: Affiris AG (Industry)
Responsible Party: Sponsor
Other Study IDs: AFF005B
Record Dates: First submitted 2011-12-16; First posted 2012-04-02 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2013-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- AFFITOPE AD03 with adjuvant
- AFFITOPE AD03 without adjuvant

SUMMARY:
This is a phase Ib follow-up study to evaluate long-term safety and tolerability of immunization with AFFITOPE AD03 applied during AFFiRiS 005A.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent signed and dated by the patient and the caregiver.
* Patients having participated in AFFiRiS 005A and received ≥1 vaccination with AFFITOPE AD03
* Availability of a partner/caregiver knowing the patient and being able to accompany the patient to the visits and being available for the telephone phone calls

Exclusion Criteria:

* Patients having received no vaccination with AFFITOPE AD03
* History of questionable compliance to visit schedule; patients not expected to complete the clinical trial

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mild to moderate Alzheimer's disease (MMSE 16 to 26)that have participated in AFF005A
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Safety/Tolerability | 52 weeks
  * Withdrawal criteria (continuation decision) Number of patients who withdraw due to AEs Reason for withdrawal
  * Number and kind (description) of AEs
  * Number and kind (description) of SAEs
  * Changes from study AFF005A in: Physical and neurological examination/ Concomitant medication/ Vital signs (blood pressure, heart rate, respiratory rate, body temperature)/ Body mass (weight)/ MRI of the brain/ ECG/ Laboratory assessment (haematology, biochemistry, coagulation, serology, APP crossreactivity and urinalysis)

SECONDARY OUTCOMES:
Clinical Efficacy | 52 weeks
  Changes from study AFF005A in:
  * CIBIC plus (Clinician's Interview-Based Impression of Change, + carer interview)
  * ADAScog (Alzheimer Disease Assessment Scale-cognitive)
  * CERAD plus (The Consortium to Establish a Registry for AD)
  * Neuropsychiatric inventory
  * Activity of daily living
  * Quality of life in patients with Alzheimer's disease
  * Investigator's global evaluation scale
  * MRI brain volumetry
Immunological | 52 weeks
  - Titre of antibodies specific for the immunizing peptide, N-terminal part of Aβ, Aβ itself, N-terminally truncated and Pyroglutamate-modified versions of Aβ, and KLH by ELlSA

CONTACTS AND LOCATIONS:
Overall Officials: Siegfried Kasper, Prof.Dr., Principal Investigator — Medical University of Vienna ,Department for Psychiatry and Psychotherapy; Dieter Volc, Prim. Dr., Principal Investigator — Studienzentrum der PROSENEX,AmbulatoriumbetriebsgesmbH an derConfraternität-Privatklinik Josefstadt
Locations (2):
- Austria (2):
  - Studienzentrum der PROSENEX, AmbulatoriumbetriebsgesmbH an derConfraternität-Privatklinik Josefstadt, Vienna
  - Medical University of Vienna, Department for Psychiatry and Psychotherapy, Vienna